CLINICAL TRIAL: NCT05679596
Title: Ketone Bodies as Therapeutic Agents to Reduce the Harmful Effects of Bed Rest on Muscle Mass and Metabolic Health in Older Adults
Brief Title: Exogenous Ketosis During Bed Rest in Older Adults
Acronym: KBR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Tyler Churchward-Venne, Principal Investigator, McGill University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 427929
Record Dates: First submitted 2022-12-12; First posted 2023-01-11 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Muscle Protein Synthesis; Muscle Atrophy; Insulin Sensitivity; Mitochondrial Function; Physical Inactivity; Cognitive Function; Muscle Strength; Functional Capacity
Keywords: Bed rest; Muscle protein synthesis; Older adults; Muscle mitochondrial function; Insulin sensitivity; Ketone bodies
MeSH Terms: conditions — Muscular Atrophy; Insulin Resistance; Sedentary Behavior | interventions — Fructose; Rapeseed Oil

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel group study design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, Investigators and Outcome Accessors will be blinded to the intervention and control drinks. The drinks will be flavor and energy matched and provided in an opaque bottle. An individual not involved with the study data collection, analysis and interpretation will be designated as a study blinder and randomizer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exogenous ketone monoester (KET) (Experimental): KET will be provided at a dose of 360 mg kg-1 body mass per serving at 2 servings per day between each main meal (ΔG®; TΔS Ltd, UK, Oxford, UK).
  Interventions: Dietary Supplement: ketone monoester (R)-3-hydroxybutyl (R)-3- hydroxybutyrate
- Energy matched control (CON) (Active Comparator): CON will be provided at a dose energy matched to the KET supplement and consist of both carbohydrate (i.e., fructose) and fat (i.e., corn and canola oil 50:50 ratio). 1/3 of the supplemental energy will come from carbohydrate while 2/3 will come from fat. We have excluded protein from the CON supplement since it is well established to influence our primary outcome measure (MPS rates). A non-caloric sweetener will also be added to the CON supplement.
  Interventions: Dietary Supplement: carbohydrate-fat placebo (fructose, corn and canola oil 50:50 ratio)

INTERVENTIONS:
Dietary Supplement: ketone monoester (R)-3-hydroxybutyl (R)-3- hydroxybutyrate — Provided twice a day between meals.
  Other Names: delta G Oxford Ketone Ester
  Arms: Exogenous ketone monoester (KET)
Dietary Supplement: carbohydrate-fat placebo (fructose, corn and canola oil 50:50 ratio) — Provided twice a day between meals.
  Arms: Energy matched control (CON)

SUMMARY:
The goal of this randomized, double-blind, parallel group interventional study is to evaluate the effect of ketone bodies on healthy older adults (65-85 y) during 5 days of bed rest. The main questions it aims to answer are:

Does supplementation of ketone bodies prevent the typical decline in muscle protein synthesis, muscle size, muscle function, insulin sensitivity, and muscle mitochondrial function that occurs in response to bed rest?

Researchers will compare ketone supplements (KET) to an energy matched control beverage (carbohydrates and fats) to see if the ketones can rescue the decline in muscle protein synthesis rates, muscle loss, muscle function, insulin sensitivity, and mitochondrial function due to 5 days of bed rest.

This may positively impact the heath of older adults subjected to bed rest.

DETAILED DESCRIPTION:
Bed rest is a common feature of many clinical environments such as hospitals and long-term care facilities. However, physical inactivity due to bed rest decreases muscle size, muscle strength, and physical performance (i.e. rising from a chair) that can lead to a reduced quality of life and a higher risk of disease and death. Eating protein-rich foods and exercising normally helps to maintain muscle size by building proteins found in muscle. However, during bed rest there is a reduction in the rate at which proteins found in muscle are made and this leads to smaller muscles. Bed rest leads to problems with blood glucose regulation and insulin resistance which can increase the risk for diabetes. Both the loss of muscle size and insulin resistance are linked to problems with parts of our cells called mitochondria. Mitochondria do a lot of important things including keeping our cells full of energy. Bed rest occurs more frequently in older adults and also negatively impacts their health more than in younger adults. Sadly, there are limited options to prevent the problems associated with bed rest. Ketone bodies are molecules that come from fat that are normally produced in the body in response to reduced carbohydrate intake (i.e. a ketogenic diet). Recently ketone supplements have become available, which increase the amount of ketone bodies in the body without the need to limit carbohydrate intake from food. Elevated ketone bodies may help protect muscle size and health during bed rest by enhancing the process of building muscle proteins, improving blood glucose regulation, and helping mitochondria work optimally.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male, and female, older adults.
* Healthy will be defined as screen by the 2020 PAR-Q+, medical screening questionnaire, GAQ, and COVID-19 symptom questionnaire patient screening.
* 'Older' will be defined as being 65-85 years of age.
* Participants are required to not engage in structured resistance training for at least 6 months prior to participation in the study.
* Participants are willing to abide by the compliance rules of this study.

Exclusion Criteria:

* Pre-menopausal females: Women must be postmenopausal having not menstruated for at least 1 year prior to study participation. Hormonal fluctuations associated with the menstrual cycle have been reported to alter protein metabolism and may influence indices of muscle protein synthesis and breakdown (69-71).
* BMI <18.5 or > 30 kg ∙ m-2.
* Self-reported regular tobacco use and vaping products.
* Self-reported illicit drug use (e.g., growth hormone, testosterone, etc.)
* Individuals who have participated in studies within the past year involving a stable isotope of 2H.
* A history of thrombosis, diagnosed with type 2 diabetes mellitus by physician or HbA1c values of > 7.0%, dementia, coronary artery disease, musculoskeletal/orthopedic disorders, and severe allergies.
* The use of medications known to modulate skeletal muscle metabolism (e.g., corticosteroids, hormone replacement therapy, non-steroidal anti-inflammatory drugs, metformin).
* The use of over-the-counter supplements (protein supplements, creatine, fish oil).
* Inability to adhere to any of the compliance rules judged by the principal investigator or medical doctor.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Changes in integrated fractional synthesis rate (%/d) in response to bed rest with and without ketone monoester (KET) supplementation. | Day 0-5 and day 5-10
  Integrative myofibrillar fractional synthesis rate will be calculated during baseline (day 0-5) and bed rest (day 5-10) phases.

SECONDARY OUTCOMES:
Changes in whole body insulin sensitivity in response to bed rest with and without ketone monoester (KET) supplementation. | Day-3 and Day 10.
  Measurements taken in the fasted state before and after bed rest. Will measure blood glucose and insulin concentration during a hyperinsulinemic-euglycemic clamp.
Changes in whole-body lean mass (kg) in response to bed rest with and without ketone monoester (KET) supplementation | Day-3 and Day 10.
  Measurements taken in the fasted state using dual-energy x-ray absorptiometry (DXA) following urinary void before and after bed rest.
Changes in leg lean mass (kg) in response to bed rest with and without ketone monoester (KET) supplementation | Day -3 and Day 10.
  Measurements taken in the fasted state using dual-energy x-ray absorptiometry (DXA) following urinary void before and after bed rest.
Changes in quadriceps muscle volume in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Measurements taken before and after bed rest via magnetic resonance imaging (MRI).
Changes in maximal voluntary isometric contraction (N/m) of the knee extensors in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Measurements taken before and after bed rest using a Biodex dynamometer.
Changes in handgrip strength (kg) in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Measurements taken before and after bed rest using a Jamar hand dynamometer.
Changes in physical performance (numerical score) as determined by short physical performance battery (SPPB) in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Measurements taken before and after bed rest
Changes in physical performance (numerical score) as determined by 5-item physical performance test in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Measurements taken before and after bed rest
Changes in cognitive status in response to bed rest with and without ketone monoester (KET) supplementation. | Day 4 and Day 9.
  NIH Toolbox Cognition Battery (computerized). Measurements taken before and after bed rest
Changes in markers of inflammation in systemic circulation in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Markers of inflammation including: IL-1 beta, NF-K beta 1, IL-6, TNF-alpha, IFNY, MIP-1 beta will be evaluated. Measurements taken before, during, and after bed rest.
Changes in muscle mRNA expression of inflammatory regulators will be assessed in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Muscle mRNA expression of NFKB1, TLR-4,IL-6, TNF-alpha, and IL-1Beta will be evaluated. Measurements taken before and after bed rest
Changes in skeletal muscle phenotype in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Muscle cross-sections immunolabeled for type I, IIa, and IIx myosin heavy chains. Measurements taken before and after bed rest.
Changes in skeletal muscle fiber size in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Muscle cross-sections analyzed for cross-sectional area.
Changes in mitochondrial content in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Via the assessment in succinate dehydrogenase activity.
Changes in mitochondrial respiration in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Assessed using standard substrate and inhibitor addition protocols in O2k high resolution Respirometer. Measurements taken before and after bed rest.
Changes in mitochondrial calcium retention capacity (marker of mitochondrial propensity to trigger apoptosis) in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Determined spectrofluorometrically using the Calcium Green probe. Measurements taken before and after bed rest.
Changes in mitochondrial reactive oxygen species (ROS) production in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Assessed using standard substrate and inhibitor addition protocols in O2k high resolution Respirometer. Measurements taken before and after bed rest.
Changes in mitochondrial time to the permeability transition pore opening (marker of mitochondrial propensity to trigger apoptosis) in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Determined spectrofluorometrically using the Calcium Green probe. Measurements taken before and after bed rest.
Changes in the phosphorylation status of anabolic signaling molecules modulating muscle protein synthesis (MPS) in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Western blotting - membranes will be probed with phospho-specific antibodies against IRS-1S527/Thr446, AktSer473, mTORSer2448, 4E-BP1Thr37/46, rpS6Ser240/244, p70S6KThr389. Measurements taken before and after bed rest.
Changes in the phosphorylation status of catabolic signaling molecules modulating muscle protein breakdown (MPB) in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Western blotting - membranes will be probed with phospho-specific antibodies against FoxO3aThr32, MuRF1, and MAFbx. Measurements taken before and after bed rest.
Blood beta-hydroxybutyrate concentrations (mmol/L) in response to bed rest with and without ketone monoester (KET) supplementation. | Day 5 and Day 10
  Measurements taken at the start and end of bed rest.
Changes in subjective pain via visual analog scale in response to bed rest with and without ketone monoester (KET) supplementation. | Day 5-10.
  Throughout the 5 day bed rest period.
Changes in muscle area in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Peripheral quantitative computed tomography (pQCT). Measurements taken before and after bed rest.
Changes in muscle density in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Peripheral quantitative computed tomography (pQCT). Measurements taken before and after bed rest.
2H enrichments in body water before and during bed rest with and without ketone monoester (KET) supplementation. | Day -1 to Day 10.
  Throughout the baseline and bed rest period.
2H-alanine enrichment in venous blood before and during bed rest with and without ketone monoester (KET) supplementation. | Day -1 to Day 10.
  Throughout the baseline and bed rest period.
Changes in resting metabolic rate (RMR) in response to bed rest with and without ketone monoester (KET) supplementation. | Day -3 and Day 10.
  Measurements taken before and after bed rest.
Physical activity level via accelerometer before bed rest. | Day 0-4.
  Throughout the baseline period
Changes in sleep disturbance (numerical score) during bed rest with and without ketone monoester (KET) supplementation. | Day 5-10.
  Via Patient-Reported Outcomes Measurement Information System (PROMIS) Short form 8a. Measured throughout the 5 day bed rest period.
Changes in sleep quality (numerical score) during bed rest with and without ketone monoester (KET) supplementation. | Day 5-10.
  Via Pittsburgh Sleep Quality Index (PSQI). Measured throughout the 5 day bed rest period.
Average habitual dietary intake assessed using Keenoa for 3 days (a food tracker application). | Measured before bed rest.
  Dietary intake will be assessed for total energy (kcals) and macronutrient (protein, carbohydrate, and fat consumption; g) intake.
Changes in Thigh Absolute Synthetic Rate (ASR) in response to bed rest with and without ketone monoester (KET) supplementation. | Day 0-5 and day 5-10
  Changes in Thigh Absolute Synthetic Rate (ASR) will be calculated during baseline (day 0-5) and bed rest (day 5-10) phases.
Changes in Thigh Absolute Protein Breakdown Rate (ABR) in response to bed rest with and without ketone monoester (KET) supplementation. | Day 0-5 and day 5-10
  Changes in Thigh Absolute Protein Breakdown Rate (ABR) will be calculated during baseline (day 0-5) and bed rest (day 5-10) phases.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler A Churchward-Venne, PhD, Principal Investigator — McGill University
Locations (1):
- Research Institute - McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No